CLINICAL TRIAL: NCT05431972
Title: Efficacy and Safety of Cardea SOLOTM for Paroxysmal Atrial Fibrillation Diagnosis in ESUS Patients With Left Atrial Enlargement: Prospective, Multi-center, Open-label, Randomized, Controlled, Investigator-Initiated Trial
Brief Title: Cardea SOLOTM for Paroxysmal Atrial Fibrillation Diagnosis in ESUS Patients With Left Atrial Enlargement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Bum Joon Kim, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SOLO-ESUS
Record Dates: First submitted 2022-06-17; First posted 2022-06-24 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Embolic Stroke of Undetermined Source
Keywords: Embolic stroke of undetermined source; left ventricle enlargement; paroxysmal atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Electrocardiography

STUDY DESIGN:
Intervention Model Description: Prospective, Multi-center, Open-label, Randomized, Controlled, Investigator-Initiated Trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cardea SOLO (Experimental): for 7 day holter monitor (patch type)
  Interventions: Device: Cardea SOLO
- 12 Lead EKG (Active Comparator): (traditional EKG for under 2 minutes)
  Interventions: Device: 12 Lead EKG

INTERVENTIONS:
Device: Cardea SOLO — Neurologist cardiac rhythm translation with 12 lead EKG versus Cardea SOLO
  Arms: Cardea SOLO
Device: 12 Lead EKG — Neurologist cardiac rhythm translation with 12 lead EKG versus Cardea SOLO
  Arms: 12 Lead EKG

SUMMARY:
The aim of the study is to evaluate the efficacy and safety of the Cardea SOLO Compared to 12 lead EKG for Paroxysmal Atrial Fibrillation Diagnosis in ESUS patients with Left Atrial Enlargement.

DETAILED DESCRIPTION:
The Prospective, Multi-center, Open-label, Randomized, Controlled, Investigator-Initiated Trial will be started on June 2022. Randomized patients in two arms will receive Cardea SOLO or 12 lead EKG respectively. Cardea SOLO received patients will keep it for 7 days. 12 lead EKG received patients will discharge home. After 7 days, Results of Cardea SOLO auto reading will be evaluated by dependent committee including cardiologist.

ELIGIBILITY:
Inclusion Criteria:

Inclusion NO. 3 or 4 must be satisfied, and No. 2, 5 and 6 must be satisfied.

2. On the Screening date, Stroke onset date is not over 60 days.

3. ESUS Diagnosis : all of a~e must be satisfied.

* a. Ischemic stroke detected by CT or MRI that is not lacunar
* b. A person without arteriosclerosis which causes at least 50% stenosis of the intracranial/external arteries supplied to the ischemic site
* c. During continuous monitoring or halter monitoring In the stroke intensive care unit, Person without atrial fibrillation and persistent atrial fibrillation
* d. When checked the Transthoracic echocardiography, No major risk cardioembolic source of embolism. (ex. Myocardial infarction within 4 weeks, mitral stenosis, artificial heart valve and so on)
* e. NO other specific cause of stroke identified(et, arteritis, dissection and drug abuse)

  4. cardioembolism is classified by TOAST classification.

  5. Left ventricle Enlargement(male >40mm, female >38mm, LAVI >35ml/m2

  6. Voluntarily sign the consent form

Exclusion Criteria:

1. Transient cerebral ischemic attack
2. Active cancer
3. Heart embolism, stroke of major heart embolism, stroke high-risk disease
4. Left atrial thrombus
5. Left ventricular thrombus
6. Sick sinus syndrome
7. Myocardiac infarction in 1 month
8. Rheumatic left atrioventricular valve or aortic valve disease
9. Artificial heart valve
10. Myocardiac infarction (EF<28%)
11. Congestive heart failure (EF<30%)
12. Dilated cardiomyopathy
13. Nonbacterial thrombotic endocarditis
14. Endocarditis
15. Intracardiac mass
16. Atrial fibrillation
17. Restriction for echocardiography (obesity, lung disease etc)
18. High risk PFO
19. Patch apply difficulty(skin allergy, ulticaria, atopic dermatitis, hyperhidrosis)
20. Implant cardiac pacemaker
21. Life-threatening arrhythmia
22. Radiation therapy or MRI scan
23. Restriction for Cardia SOLO attachment
24. The person who investigator judged unsuitable for the trial

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2024-09-13 (Actual)

PRIMARY OUTCOMES:
Patients number with AF over 30 seconds of cardea SOLO / with AF with 1 time of 12 lead EKG | 30 seconds
  cardea SOLO and 12 lead EKG is different

SECONDARY OUTCOMES:
AF burden(F) | 1 week
  cardea SOLO and 12 lead EKG is different
Number of other dysrhythmia | 1 week
  cardea SOLO and 12 lead EKG is different

CONTACTS AND LOCATIONS:
Locations (1):
- BumJoon Kim, Seoul, South Korea